CLINICAL TRIAL: NCT05526768
Title: Evaluation of a Novel Remote Vital Sign Monitor Compared to Traditional Inpatient Monitoring in Cardiac Shunt-Dependent Children
Brief Title: Evaluation of VITLS Compared to Traditional Inpatient Monitoring in Cardiac Shunt-Dependent Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Southwest National Pediatric Device Innovation Consortium (SWPDC) (Unknown)
Responsible Party: Principal Investigator, Pamela Carol Petersen, Assistant Professor of Pediatric Critical Care Medicine, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H-46463
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Congenital Heart Disease; Desaturation of Blood
Keywords: remote monitoring; pulse oximeter; cardiac shunt dependent; Tego; VITLS
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Masking Description: The providers caring for the participating patients will be blinded to the data being collected by the remote monitoring system and no patient care decisions will be made based on the remote monitoring system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VITLS Device (Experimental): The remote monitoring device (VITLS) will be placed onto the chest of consented patients in a manner that will not interfere with standard in-patient monitoring devices. Subjects will simultaneously be monitored with conventional inpatient methods per the unit routine. The providers caring for participating patients will be blinded to the data being collected by the remote monitoring system and no patient care decisions will be made based on the remote monitoring system. The remote monitoring device will automatically monitor and store the data for each subject by subject ID number. Once at least 6, but up to 72 hours of data have been recorded, the investigational device will be removed. Researchers will then retrospectively obtain the corresponding data from the current standard of care inpatient monitoring devices.
  Interventions: Device: VITLS Device

INTERVENTIONS:
Device: VITLS Device — VITLS remote vital sign monitoring device will be applied to consented patients so data obtained by the device can be compared to data obtained by traditional inpatient hospital monitoring devices.

SUMMARY:
We are seeing how well a remote monitoring device that looks like a sticker placed on the chest, under the arm can monitor a child's vital signs including oxygen levels compared to the way that we usually get these measurements. The goal of this study is to see if the new sticker can be used for monitoring patients with cardiac shunt dependent heart conditions from home once they are discharged home. Participating children will be monitored for 6-72 hours with the new sticker in addition to his/her usual hospital monitors so the new sticker device can be compared to our hospital monitors.

DETAILED DESCRIPTION:
Children with congenital heart disease who are cardiac shunt dependent are at increased risk for physiologic decompensation compared to non-shunt dependent children. This can lead to prolonged hospitalizations to facilitate careful vital sign monitoring to detect signs of deterioration early. While home monitoring programs have shown promise in this population, there is currently a shortage of pediatric specific remote monitoring devices that seamlessly provide vital sign results to caregivers and the healthcare team.

Over the past few years, home monitoring programs utilizing portable pulse oximetry to monitor oxygen saturation at home have reported improved survival in infants with single ventricle (cardiac shunt dependent) heart disease. Monitoring vital signs in cardiac shunt-dependent children presents challenges as most pulse oximeters are designed to monitor saturation levels greater than 85% SpO2 and shunt dependent children have baseline saturations closer to 75-85% SpO2. Additionally, traditional pulse oximetry probes are connected to a stationary monitor by leads of varying lengths. Children can easily remove these leads, thereby requiring frequent repositioning of the pulse oximeter. Additional limitations to current technology include inaccurate measurements due to motion artifact, need for frequent probe changes, parental requirement to log and interpret results, and the machines' lack of recording ability. An ideal monitor would be one that has continuous monitoring and recording features and provides feedback to the health care team in real time.

This study aims to evaluate a potential solution to some of the problems faced in home monitoring of cardiac shunt-dependent children. The proposed study device continuously measures pulse oximetry, heart rate, respiratory rate and temperature via a wireless probe that is placed on the child's chest. The device wirelessly transmits and stores the vital sign data continuously and can be accessed by authorized medical providers and the patient's caregivers at all times. The goal of this pilot study is to measure how the study device performs in comparison to standard-of-care hospital monitoring in the patients of interest.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac shunt-dependent patients aged 0-1 year old located in the Texas Children's Hospital Cardiac Intensive Care Unit (CVICU)

Exclusion Criteria:

* Presence of any implanted metal or electronic medical devices present in the chest (i.e. pace makers)
* Allergy to medical grade (latexfree) adhesive
* Any congenital or acquired desquamating skin condition (e.g., staphylococcal scalded skin syndrome, Stevens-Johnson syndrome, toxic epidermal necrolysis)
* Any other medical condition which, in the opinion of the Investigator, could affect the participant's health during trial participation or could compromise his/her ability to participate in the trial.
* In the opinion of the investigator, the participant and his/her parent(s) or legal guardian(s) is not reliable for participation in the trial.
* Parental language of comfort is not English or Spanish.
* Parents do not consent for study inclusion.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of pulse oximetry | 6-72 hours
  Evaluate the VITLS device's ability to accurately measure pulse oximetry compared to conventional inpatient wall-connected methods in cardiac shunt-dependent children.

SECONDARY OUTCOMES:
Evaluate the ability of VITLS to detect clinically significant SpO2 vital sign events compared to conventional inpatient methods. | 6-72 hours
  Clinically significant SpO2 vital sign events are defined as SpO2 less than 75% or SpO2 greater than 90% sustained for 1 minute.
Evaluate the ability of VITLS to detect clinically significant Heart Rate vital sign events compared to conventional inpatient methods. | 6-72 hours
  Clinically significant vital sign events are defined as heart rate less than 100 bpm or heart rate greater than 180 bpm sustained for 1 minute.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela C Petersen, MD, Principal Investigator — Texas Children's Hospital/Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No